CLINICAL TRIAL: NCT00269204
Title: A Worldwide, Multicenter, Double-Blind, Randomized, Parallel, Placebo-Controlled Study to Evaluate the Lipid-Altering Efficacy, Safety and Tolerability of MK0524A in Patients With Primary Hypercholesterolemia or Mixed Hyperlipidemia
Brief Title: Lipid Efficacy/Tolerability Study (0524A-020)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0524A-020; MK0524A-020; 2005_095
Record Dates: First submitted 2005-12-21; First posted 2005-12-23 (Estimated); Last update posted 2015-07-27 (Estimated); Status verified 2015-07

CONDITIONS: Primary Hypercholesterolaemia; Mixed Hyperlipidaemia
MeSH Terms: conditions — Hyperlipoproteinemia Type II | interventions — Niacin; MK-0524

STUDY DESIGN:
Who Masked: Participant, Investigator

INTERVENTIONS:
Drug: niacin (+) laropiprant — Duration of Treatment - 24 weeks
  Other Names: MK0524A
Drug: ER-niacin — Duration of Treatment - 24 weeks

SUMMARY:
A 28-week clinical trial in patients with primary hypercholesterolemia or mixed hyperlipidemia to study the effects of MK0524A on lipids and tolerability. There will be 9 scheduled clinic visits, and 3 treatment groups. A patient can be randomly assigned to 1 of the 3 treatment groups.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 to 85 years of age with Primary Hypercholesterolemia or Mixed Hyperlipidemia with LDL-C below 100 mg/dL for high risk patients (patients with Coronary Artery Disease (CHD).
* Have medical conditions considered to be CHD equivalent).
* LDL-C below 130 mg/dL for patients with multiple risk factors.
* LDL-C between 130 and 190 mg/dL for patients with low risk and Triglycerides </= to 350 mg/dL.

Exclusion Criteria:

* A condition which, in the opinion of the investigator, might pose a risk to the patient or interfere with participating in the study, patients < 20% compliance, patients with chronic medical conditions, patients with unstable doses of medications.
* Pregnant or lactating women, or women intending to become pregnant are excluded.
* Patient with diabetes mellitus that is poorly controlled, newly diagnosed, has recently experienced repeated hypoglycemia or unstable glycemic control, or is taking new or recently adjusted antidiabetic pharmacotherapy (with the exception of +/- 10 units of insulin).
* Patients with the following conditions: chronic heart failure, uncontrolled/unstable cardiac arrhythmias, unstable hypertension, active or chronic hepatobiliary or hepatic disease, HIV positive, gout (within 1 year).

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1620 (Actual)
Dates: Start 2005-12; Primary Completion 2006-12 (Actual); Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
Reductions of LDL-C concentrations at 24 weeks and better tolerability | at 24 weeks

SECONDARY OUTCOMES:
Elevations in HDL-C concentrations at 24 weeks | at 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Background] Baron JA, Sandler RS, Bresalier RS, Quan H, Riddell R, Lanas A, Bolognese JA, Oxenius B, Horgan K, Loftus S, Morton DG; APPROVe Trial Investigators. A randomized trial of rofecoxib for the chemoprevention of colorectal adenomas. Gastroenterology. 2006 Dec;131(6):1674-82. doi: 10.1053/j.gastro.2006.08.079. Epub 2006 Sep 1. PMID 17087947
- [Background] Maccubbin D, Bays HE, Olsson AG, Elinoff V, Elis A, Mitchel Y, Sirah W, Betteridge A, Reyes R, Yu Q, Kuznetsova O, Sisk CM, Pasternak RC, Paolini JF. Lipid-modifying efficacy and tolerability of extended-release niacin/laropiprant in patients with primary hypercholesterolaemia or mixed dyslipidaemia. Int J Clin Pract. 2008 Dec;62(12):1959-70. doi: 10.1111/j.1742-1241.2008.01938.x. PMID 19166443
- [Background] Bays HE, Maccubbin D, Meehan AG, Kuznetsova O, Mitchel YB, Paolini JF. Blood pressure-lowering effects of extended-release niacin alone and extended-release niacin/laropiprant combination: a post hoc analysis of a 24-week, placebo-controlled trial in dyslipidemic patients. Clin Ther. 2009 Jan;31(1):115-22. doi: 10.1016/j.clinthera.2009.01.010. PMID 19243712
- [Derived] Rao M, Steffes M, Bostom A, Ix JH. Effect of niacin on FGF23 concentration in chronic kidney disease. Am J Nephrol. 2014;39(6):484-90. doi: 10.1159/000362424. Epub 2014 May 20. PMID 24854458
- [Derived] Bays HE, Shah A, Lin J, Sisk CM, Dong Q, Maccubbin D. Consistency of extended-release niacin/laropiprant effects on Lp(a), ApoB, non-HDL-C, Apo A1, and ApoB/ApoA1 ratio across patient subgroups. Am J Cardiovasc Drugs. 2012 Jun 1;12(3):197-206. doi: 10.2165/11631530-000000000-00000. PMID 22500948
- [Derived] Bays H, Shah A, Dong Q, McCrary Sisk C, Maccubbin D. Extended-release niacin/laropiprant lipid-altering consistency across patient subgroups. Int J Clin Pract. 2011 Apr;65(4):436-45. doi: 10.1111/j.1742-1241.2010.02620.x. PMID 21401833